CLINICAL TRIAL: NCT00730782
Title: Assessment of the Safety and Immunogenicity of Three Formulations of the Recombinant Pichia Pastoris Apical Membrane Antigen 1 (PfAMA-1-FVO[25-545]), Blood-Stage Malaria Vaccine in Healthy Dutch Adult Volunteers : a Phase 1, Single- Blind, Randomised, Dose-Escalating, Unicentre Trial
Brief Title: Assessment of Three Formulations of the Candidate Vaccine AMA 1 in Healthy Dutch Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: European Vaccine Initiative (Other)
Collaborators: Radboud University Medical Center (Other); Biomedical Primate Research Centre (Other); GlaxoSmithKline (Industry); Seppic (Industry)
Responsible Party: Prof. Dr. R.W. Sauerwein, Radboud University Nijmegen Medical Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AMA-1_1_03; EUDRACT No 2005-00232-24
Record Dates: First submitted 2008-08-06; First posted 2008-08-08 (Estimated); Last update posted 2008-08-08 (Estimated); Status verified 2008-08

CONDITIONS: Plasmodium Falciparum Malaria
MeSH Terms: conditions — Malaria, Falciparum

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): The experimental vaccine PfAMA1 formulated in Alhydrogel
  Interventions: Biological: PfAMA-1-FVO[25-545]
- 2 (Active Comparator): The experimental vaccine PfAMA1 formulated in Montanide ISA720
  Interventions: Biological: PfAMA-1-FVO[25-545]
- 3 (Active Comparator): The experimental vaccine PfAMA1 formulated in ASO2A
  Interventions: Biological: PfAMA-1-FVO[25-545]

INTERVENTIONS:
Biological: PfAMA-1-FVO[25-545] — Subcutaneous vaccination of 0.5ml of two dosage 10 and 50ug PfAMA1

SUMMARY:
The objective of this study was to evaluate the safety of a candidate malaria vaccine (PfAMA-1) at 3 doses given at monthly intervals of 2 different dosages of AMA-1 (10 μg or 50 μg ) adjuvanted either with alum hydroxide or AS02A or Montanide ISA 720 in healthy adults not previously exposed to the parasite Plasmodium falciparum.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 and < 45 years healthy volunteers.
* General good health based on history and clinical examination.
* All volunteers have to sign the informed consent form.
* Negative pregnancy test.
* Use of adequate contraception for females up to three months after the third injection (D140).
* Reachable by phone during the whole study period (18 months).

Exclusion Criteria:

* History of malaria or residence in malaria endemic areas within the past six months.
* Positive serology for malaria antigen PfAMA-1
* Previously participated in any malaria vaccine study
* Symptoms, physical signs and laboratory values suggestive of systemic disorders, including renal, hepatic, cardiovascular, pulmonary, skin, immunodeficiency, psychiatric and other conditions, which could interfere with the interpretation of the study results or compromise the health of the volunteers.
* Any laboratory abnormalities on screened blood samples beyond the normal range, as defined at UMC St Radboud. Positive HIV, HBV or HCV tests.
* Volunteers should not be enrolled in any other clinical trial during the whole trial period.
* Volunteers should not receive chronic medication, especially immunosuppressive agents (steroids, immunomodulating or immunosuppressive drugs) during the three months preceding the screening visit or during the study period.
* Pregnant or lactating women.
* Volunteers unable to give written informed consent.
* Volunteers unable to be closely followed for social, geographic or psychological reasons.
* Previous history of drug or alcohol abuse interfering with normal social function during a period of one year prior to enrollment in the study.
* Volunteers should not perform exercise four hours before blood draw and should not donate blood for non study-related purposes during the entire duration of the study.
* Known hypersensitivity to any of the vaccine components (adjuvant or peptide).
* Volunteers are not allowed to receive any vaccination or gammaglobulin during a period three months prior to the first immunization and up to six months after the 3rd immunization. If a vaccination is necessary during this period, the volunteer will be withdrawn from the study.
* Volunteers are not allowed to travel to malaria endemic countries during the study period.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2005-11; Primary Completion 2007-09 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Local and systemic reactogenicity | Day 0-14 after each vaccination

SECONDARY OUTCOMES:
Biological Safety | 28 days after each vaccination
Humoral and Cellular immunogenicity | until 365 days after the first immunisation

CONTACTS AND LOCATIONS:
Overall Officials: Robert Sauerwein, Prof. MD, Principal Investigator — Radboud University Medical Center
Locations (2):
- Netherlands (2):
  - Radboud University Nijmegen Medical Centre, Nijmegen
  - Biomedical Primate Research Centre, Rijswijk

REFERENCES:
- [Derived] Remarque EJ, Roestenberg M, Younis S, Walraven V, van der Werff N, Faber BW, Leroy O, Sauerwein R, Kocken CH, Thomas AW. Humoral immune responses to a single allele PfAMA1 vaccine in healthy malaria-naive adults. PLoS One. 2012;7(6):e38898. doi: 10.1371/journal.pone.0038898. Epub 2012 Jun 29. PMID 22768052
- [Derived] Roestenberg M, Remarque E, de Jonge E, Hermsen R, Blythman H, Leroy O, Imoukhuede E, Jepsen S, Ofori-Anyinam O, Faber B, Kocken CH, Arnold M, Walraven V, Teelen K, Roeffen W, de Mast Q, Ballou WR, Cohen J, Dubois MC, Ascarateil S, van der Ven A, Thomas A, Sauerwein R. Safety and immunogenicity of a recombinant Plasmodium falciparum AMA1 malaria vaccine adjuvanted with Alhydrogel, Montanide ISA 720 or AS02. PLoS One. 2008;3(12):e3960. doi: 10.1371/journal.pone.0003960. Epub 2008 Dec 18. PMID 19093004